CLINICAL TRIAL: NCT03049423
Title: MRI Appearance of Injured Ligament and Tendon of the Ankle in Different Postures: Study Protocol for a Single-center, Diagnostic Clinical Trial
Brief Title: MRI Appearance of Injured Ligament and Tendon of the Ankle in Different Postures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Guobin Liu, Chief Physician, The First Hospital of Hebei Medical University
Other Study IDs: FirstHebei_002
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Magnetic Resonance Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the trial group: 30 patients with ankle ligament and tendon injury were selected in accordance with the diagnostic criteria of ankle ligament and tendon injury in the trial group. Each participant was required to undergo MRI scans in normal position and during complete plantar flexion and complete dorsiflexion.
  Interventions: Device: MRI scans
- the control group: 30 patients with normal ankle joint were selected in accordance with the diagnostic criteria of ankle ligament and tendon injury in the control group. Each participant was required to undergo MRI scans and general physical examination in normal position and during complete plantar flexion and complete dorsiflexion.
  Interventions: Diagnostic Test: MRI scans and general physical examination

INTERVENTIONS:
Device: MRI scans — 30 patients with ankle ligament and tendon injury were selected in accordance with the diagnostic criteria of ankle ligament and tendon injury in the trial group. Each participant was required to undergo MRI scans in normal position and during complete plantar flexion and complete dorsiflexion.
  Groups: the trial group
Diagnostic Test: MRI scans and general physical examination — 30 patients with normal ankle joint were selected in accordance with the diagnostic criteria of ankle ligament and tendon injury in the control group. Each participant was required to undergo MRI scans and general physical examination in normal position and during complete plantar flexion and complete dorsiflexion.
  Groups: the control group

SUMMARY:
To compare the results of multi-position MRI scans for ankle ligaments and tendons to clarify how to obtain imaging data of different ankle ligaments and define severity of injuries to calculate the rate of correct diagnosis, thereby developing a reasonable surgical treatment in clinical practice.

DETAILED DESCRIPTION:
The ankle joint is an important part of the human lower limb. It has the function of maintaining the normal standing of the human body, supporting and bearing the body weight and conducting movements. As one of the complex joints of the human body, its surrounding ligaments and tendons not only play an important protective effect on it, but also play a fixed role in the movement of the ankle to effectively prevent excessive ankle varus/valgus. Ankle fractures account for approximately 3.9% of total body fractures, ranking the first in intra-articular fractures. An ankle injury is often accompanied by intra-articular fractures and surrounding ligament rupture. With the increasing requirements for joint functions and clinical surgery, inappropriate treatment for ankle ligament injury can result in limited movement function of the ankle, and even lead to traumatic arthritis and chronic ankle instability.

X-ray examinations are routinely preferred for the diagnosis of ankle injury, which can make an accurate diagnosis of ankle dislocation and fracture. However, X-ray plain film has a low resolution for tendon and ligament lesions, which is easy to result in missed diagnosis of mild fractures, bone contusion and occult fractures, and moreover, it is difficult to fully clear the location, type and degree of ankle injury.

MRI has high definition and resolution to implement a multi-parameter multi-directional scanning. Its histopathological findings can accurately and objectively display ankle and surrounding ligament injuries and their severity. MRI is able to display the anatomic structure and severity of ligament injury of the ankle on three anatomic planes: transverse, sagittal and coronal. Sagittal MRI is a good helper for diagnosis of Achilles tendon lesion, which can clearly show the talus, posterior tibial tendon, talocalcaneal joint, Achilles tendon, subtalar joint, articulatio talonavicularis, tibiotalar joint, and the cartilage and joint cavities. Coronal MRI can clearly show structures of the peroneal joint, tibiotalar joint, and lateral malleolus, especially the articular surface between the tibia, fibula and the ankle bone as well as between the ligament fibula and the ankle bone; and meanwhile, it can display the posterior tibial ligament, posterior talofibular ligament and posterior tibial tendon. Transverse MRI well shows the tibiofibular ligament, and anterior talofibular ligament. The ankle ligament mainly consists of three parts: the lateral collateral ligament, medial collateral ligament and tibiofibular ligament. Activities of the ankle refer to flexion and extension along the sagittal plane, including plantar flexion and dorsiflexion, to play a role of supporting and bearing, movement conduction and function as a lever.

Adverse events If expected or unexpected adverse events (such as headache and nausea) during the MRI detection, the date of occurrence, type of injury and therapeutic managements will be recorded. Severe adverse events, including a requirement for immediate surgery, damage to patient's work ability, life-threatening events or death will be reported to the project manager and the institution review board within 24 hours.

Data collection, management, analysis and open access All data will be collected on a case report form, recorded electronically and saved in a dedicated computer. Continuous variables from each record will be collected for descriptive statistical analysis, to allow real-time review and identify any potential deviation.

The validity of the data will be assessed by the censor once every 6 months through a random sampling of 10% of the database. Only the researchers participating in the study will have the right to query the database that will not be modified.

Statistical analysis will be completed by professional statisticians who will responsible for a statistical report. The statistical results will be given to the project manager, who will be responsible for writing the research report.

Anonymized trial data will be released at www.figshare.com.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for ankle ligament and tendon injury
* Age 34-78 years
* Both genders
* Sign the informed consent prior to the trial

Exclusion Criteria:

* Heart, liver, kidney and other important organ diseases
* Ankle open fracture
* Old fracture of the ankle joint
* An open tendon or ligament rupture of the ankle
* Neuropsychiatric disorders (epilepsy, depression or panic disorder)
* Pregnant or lactating women
* Participate in other clinical trials over the past 3 months

Ages: 34 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Six participants from the First Affiliated Hospital of Hebei Medical University were recruitment through newspapers, public communication, hospital and public institution websites. The participants gave written informed consent prior to participation in the trial.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of MRI scan for ligament and tendon injury of the ankle | during the MRI scan
  The sensitivity (true positive rate) is defined as the percentage of actual patients who are correctly diagnosed with a disease. A higher sensitivity indicates a higher rate of correct diagnosis.

SECONDARY OUTCOMES:
The specificity of MRI scan for ligament and tendon injury of the anklethe ankle | during the MRI scan
  The specificity (true negative rate) is defined as the percentage of disease-free patients who are correctly diagnosed with no disease. A higher specificity indicates a higher rate of correct diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Guobin Liu, Master, Principal Investigator — The First Affiliated Hospital of Hebei Medical University

IPD SHARING:
Plan to Share IPD: Undecided